CLINICAL TRIAL: NCT03182335
Title: An Assessment of Vasoactive Medication Dose in Mechanically Ventilated Patients Undergoing Daily Sedation Awakening Trial (SAT)
Brief Title: Vasopressor SAT Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1532
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Low Blood Pressure; Delirium; Critical Illness
MeSH Terms: conditions — Hypotension; Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mechanical Ventilation (MV) with vasoactive infusions: adult ICU patients who are mechanically ventilated with sedative infusion and/or analgesic infusion and also requiring vasoactive drug infusions for the treatment of shock. Patients will be excluded if receiving dexmedetomidine as sedative.
  Interventions: Other: sedation awakening trial

INTERVENTIONS:
Other: sedation awakening trial — vital signs and delirium assessment (CAM-ICU) at baseline then following routine sedation awakening trial. Patient will thus serve as their own control for these interventions
  Other Names: SAT

SUMMARY:
To assess the impact of daily awakening from sedation on the amount of vasoactive medication required in the ICU. The hypothesis of this proposal is that the amount of vasoactive drug required to maintain an adequate mean arterial blood pressure will be reduced during a daily awakening from sedation.

DETAILED DESCRIPTION:
This observational study will compare mean arterial pressure and vasoactive drug dose recorded at two time points:

1. prior to awakening from sedation
2. during the awakening from sedation trial The vasoactive infusion will be titrated to a mean arterial pressure as determined by the medical team prior to study enrollment. Each enrolled patient will have measurements taken only on the first day of enrollment. Enrolled subjects will also have a delirium assessment using the CAM-ICU tool before the awakening from sedation trial and during the awakening from sedation trial.

ELIGIBILITY:
Inclusion Criteria:

* requiring Mechanical ventilation through an endotracheal tube with infusion of sedative or analgesic agent for comfort
* requiring vasoactive drug via central venous catheter for the treatment of shock

Exclusion Criteria:

* patients receiving Dexmedetomidine as sedative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-04-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
change in vasoactive drug dose | baseline thru study completion on average < 4 hrs
  mcg/kg/min baseline dose and nadir dose

SECONDARY OUTCOMES:
change in mean arterial blood pressure | baseline thru study completion on average <4 hrs
  mm Hg
change in prevalence of ICU delirium | baseline thru study completion on average <4hrs
  CAM ICU score

CONTACTS AND LOCATIONS:
Overall Officials: John Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided